CLINICAL TRIAL: NCT00489138
Title: Prospective, Open-label Study of Pharmacokinetics of Ertapenem in the Muscle Using Microdialysis in Mechanically Ventilated Intensive Care Unit Patients, Treated or Not by Norepinephrine
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006/24
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: To Assess the Tissular and Plasma Kinetics of Ertapenem
MeSH Terms: interventions — Ertapenem

ARMS (2):
- 1 (Experimental): Noradrenalin infusion
  Interventions: Drug: Ertapenem
- 2 (No Intervention): No adrenalin infusion

INTERVENTIONS:
Drug: Ertapenem — 1g a day by drip of 30 min
  Arms: 1

SUMMARY:
Goal of study:

To assess the tissular and plasma kinetics of ertapenem;

To determine the optimal dosages in the patients according to norepinephrine administration:

* to assess muscular diffusion of free form of ertapenem after administration to mechanically ventilated patients requiring such a treatment. The patients are included in the groups "with norepinephrine" or "without norepinephrine" according to their hemodynamic status.
* to assess the plasma pharmacokinetics of ertapenem in mechanically ventilated patients treated or not by norepinephrine.

Open-label, prospective study performed in a single ICU (16 beds) of a tertiary hospital (700 beds).

ELIGIBILITY:
Inclusion Criteria:

* 18 years and more
* negative pregnancy test
* HIV/HBV, HCV negative tests
* Mechanical ventilation with pneumonia or intraabdominal infection requiring ertapenem

Exclusion Criteria:

* refractory septic shock requiring use of additional catecholamines
* patients with positives tests for HIV, HBV, HCV
* pregnant females
* allergic insufficiency
* hemodiafiltration
* contraindication to microdialysis catheter set-up
* severe arteritis of lower extremities
* treatment with vasodilatators
* prior history of aorto-iliac shunt
* involvement in a clinical trial in the last three months
* exclusion from national records
* non affiliated to "securité sociale"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
assess the tissular and plasma kinetics of ertapenem | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ioanna BOYADJIEV, PH, Principal Investigator — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Département d'Anesthésie-Réanimation - CHU NORD, Marseille, France

REFERENCES:
- [Derived] Boyadjiev I, Boulamery A, Simon N, Martin C, Bruguerolle B, Leone M. Penetration of ertapenem into muscle measured by in vivo microdialysis in mechanically ventilated patients. Antimicrob Agents Chemother. 2011 Jul;55(7):3573-5. doi: 10.1128/AAC.00180-11. Epub 2011 May 16. PMID 21576440